CLINICAL TRIAL: NCT02729714
Title: A Randomized, Double-Blind, Placebo-Controlled Pilot Study of Suvorexant for Insomnia in Parkinson Disease
Brief Title: A Pilot Study of Suvorexant for Insomnia in Parkinson Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Burdick, Daniel, M.D. (Individual)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Daniel Burdick, MD, Principal Investigator, Burdick, Daniel, M.D.
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: DJB-2015-01
Record Dates: First submitted 2016-01-26; First posted 2016-04-06 (Estimated); Results first posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-07

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — suvorexant; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Suvorexant or Placebo (Active Comparator): 10 Suvorexant or Placebo mg orally at bedtime with an optional up-titration to 15 mg Suvorexant or Placebo orally at bedtime after 2 weeks. The first treatment period will be 4 weeks. Subjects will be randomized 1;1 to receive Suvorexant or matching placebo. Followed by a 2 week washout period with placebo. Subjects will then be crossed over into the alternate treatment group. Subjects on active treatment for period 1 will be switched to placebo, those on placebo in period 1 will switch to Suvorexant
  Interventions: Drug: Suvorexant; Drug: Placebo
- Placebo or Suvorexant (Placebo Comparator): First treatment period will be 4 week which subjects will be randomized 1;1 with either Suvorexant or placebo. Followed by 2 week washout period with placebo. Subjects will then be crossed over into the alternate treatment group. Subjects on active treatment for period 1 will be switched to placebo, those on placebo in period 1 will switch to Suvorexant.
  Interventions: Drug: Suvorexant; Drug: Placebo

INTERVENTIONS:
Drug: Suvorexant — 10 mg Suvorexant or matching Placebo orally at bedtime with optional up-titration to 15 mg Suvorexant or matching Placebo orally at bedtime after 2 weeks.
  Other Names: Belsomra
Drug: Placebo — 10 mg Suvorexant or matching Placebo orally at bedtime with optional up-titration to 15 mg Suvorexant or matching Placebo orally at bedtime after 2 weeks.
  Other Names: Sugar Pill

SUMMARY:
The purpose of this study is to see if the study drug, suvorexant, is safe and effective in treating symptoms of insomnia in people with Parkinson's Disease. It is anticipated that a total of 20 subjects, 30 to 80 years of age, with Parkinson's Disease and symptoms of insomnia will participate in the study at this site

DETAILED DESCRIPTION:
The proposed study is a randomized, double-blind, placebo-controlled, cross-over trial to assess the safety, tolerability, and efficacy of suvorexant specifically in a cohort of 20 Parkinson's Disease patients between the ages of 30 and 80 (inclusive) who have a complaint of insomnia. After informed consent is given, potential subjects will be screened to ensure they meet eligibility criteria. This will include an overnight polysomnogram, which will serve both as a baseline and a screening polysomnogram. Active drug will be suvorexant 10 mg orally at bed time with an optional up-titration to 15 mg orally at bedtime after 2 weeks. The first treatment period will be 4 weeks long, in which subjects will be randomized 1:1 to receive active drug or matching placebo. At the end of treatment period 1, subjects will undergo efficacy assessment with repeat polysomnogram and clinical scales. This will be followed by a 2-week washout period with placebo; this period only will be single-blinded, as subjects only will be blinded to treatment. Subjects will then be crossed over into the alternate treatment group, which will once again be double-blinded; those on active treatment for period 1 will be switched to placebo, and those on placebo in period 1 will be switched to active treatment. Treatment period 2 will also be 4 weeks long, and at the end of this, subjects will undergo final assessment with polysomnogram and clinical scales.

ELIGIBILITY:
Inclusion Criteria:

* Has signed and dated an Institutional Review Board-approved informed consent form before any protocol-specific screening procedures are performed;
* Has a diagnosis of Parkinson disease according to the United Kingdom Parkinson Disease Society Brain Bank Criteria;
* Has a modified Hoehn and Yahr Stage of 1-3, inclusive;
* Is aged 30-80 years old, inclusive;
* Has had no change in Parkinson's Disease medications during the 4 weeks preceding screening, with no dose changes during the study, except that as needed doses of carbidopa/levodopa will be allowed to address periodic worsening of parkinsonian symptoms;
* Is willing and able to complete polysomnogram;
* Is subject willing and able to limit alcohol use to 1 alcoholic drink per day during the study period and abstain from alcohol for 6 hours prior to each study-related polysomnogram?
* Is subject willing and able to abstain from caffeine and marijuana for 6 hours prior to and during each study-related polysomnogram
* Is subject willing and able to abstain from products containing nicotine during each study-related polysomnogram?
* Has Insomnia Disorder defined by diagnostic criteria published in the Diagnostic and Statistical Manual of Mental Disorders, 5th edition; namely, subject report of all of the following:

  * One of the following: difficulty initiating sleep; difficulty maintaining sleep; or early morning waking;
  * Sleep disturbance causes clinically significant distress or impairment in social, occupational, educational, academic, behavioral, or other important areas of functioning;
  * Sleep difficulty has occurred on 3 or more nights per week;
  * Sleep difficulty has been present for at least the past 3 months;
  * Sleep difficulty occurs despite adequate opportunity for sleep;
  * Insomnia is not explained by another sleep disorder;
  * Insomnia is not attributable to physiological effects of a consumed substance;
* On screening polysomnogram, has a latency to persistent sleep > 20 minutes OR total wakefulness after sleep onset > 45 minutes;
* May use other medications that could influence sleep, other than those specifically prohibited, as long as the dose is stable for 4 weeks preceding screening, with no dose changes during the study; and
* Has valid health insurance coverage at the time of study enrollment and expects this coverage to remain valid for the duration of the study period.

Exclusion Criteria:

* Is a woman who is breast-feeding, pregnant, or has the potential to become pregnant during the course of the study (fertile and unwilling/unable to use effective contraceptive measures);
* Does subject have an implanted deep brain stimulator?
* Has a history of narcolepsy;
* Has a diagnosis of severe chronic obstructive pulmonary disease, defined by forced expiratory volume in 1 second < 50% of predicted on most recent available pulmonary function test (a pulmonary function test is not required if the subject has never been diagnosed with chronic obstructive pulmonary disease);
* Has a history of severe obstructive sleep apnea or evidence of severe obstructive sleep apnea on screening polysomnogram, with severe obstructive sleep apnea defined as having an apnea-hypopnea index > 30;
* Is concurrently using other central nervous system depressants, including alcohol, except that one alcoholic drink per day will be allowed for those with normal hepatic function provided the drink is consumed at least 2 hours prior to or 8 hours after taking the study drug, and no alcohol will be permitted for 24 hours before polysomnogram visits;
* Is concurrently using digoxin;
* Is concurrently using any moderate or strong inhibitor of cytochrome P450 3A;
* Is concurrently using any strong inducer of cytochrome P450 3A;
* Has evidence at screening of severe hepatic impairment as defined by a Child-Pugh score > 10;
* Has evidence at screening of severe cognitive impairment as defined by a Montreal Cognitive Assessment score < 15, or has cognitive impairment that in the opinion of the investigator would prevent completion of study procedures or the ability to provide informed consent.
* Has evidence at screening of suicidal ideation in the past 6 months as defined by a positive response to any one of Questions 2-5 on the Columbia Suicide Severity Rating Scale or of a lifetime history of suicidal behavior as defined by any positive response to the suicidal behavior section of the Columbia Suicide Severity Rating Scale.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2022-04 (Actual); Study Completion 2022-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Burdick, MD, Principal Investigator — Booth Gardner Parkinson's Care Center
Locations (1):
- Evergreenhealth Booth Gardner Parkinsons Care Center, Kirkland, Washington, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Suvorexant Then Placebo: 10 Suvorexant or Placebo mg orally at bedtime with an optional up-titration to 15 mg Suvorexant or Placebo orally at bedtime after 2 weeks. The first treatment period will be 4 weeks. In this group, subjects were randomized 1:1 to receive Suvorexant in the first period. Following a 2 week washout period with placebo, subjects in this group were crossed over into the placebo group for the second treatment period, also 4 weeks.
- Placebo Then Suvorexant: 10 Suvorexant or Placebo mg orally at bedtime with an optional up-titration to 15 mg Suvorexant or Placebo orally at bedtime after 2 weeks. The first treatment period will be 4 weeks. In this group, subjects were randomized 1:1 to receive Placebo in the first period. Following a 2 week washout period with placebo, subjects in this group were crossed over into the suvorexant group for the second treatment period, also 4 weeks.
Period: Treatment Period 1 (4 Weeks)
Arm/Group | Suvorexant Then Placebo | Placebo Then Suvorexant
Started | 11 | 10
Completed | 11 | 10
Not Completed | 0 | 0
Period: Washout Period (2 Weeks)
Arm/Group | Suvorexant Then Placebo | Placebo Then Suvorexant
Started | 11 | 10
Completed | 11 | 9
Not Completed | 0 | 1
Period: Treatment Period 2 (4 Weeks)
Arm/Group | Suvorexant Then Placebo | Placebo Then Suvorexant
Started | 11 | 9
Completed | 11 | 8
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Suvorexant Then Placebo | Placebo Then Suvorexant | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.1 (9.4) | 55.9 (5.6) | 60.2 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 6
  Male | 6 | 9 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 9 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 10 | 21
Years since diagnosis of Parkinson disease [Mean (Standard Deviation); unit: years] | 3.4 (3.0) | 3.9 (2.3) | 3.7 (2.7)
Levodopa-Equivalent Daily Dose [Mean (Standard Deviation); unit: mg] | 687.8 (336.0) | 676.9 (213.6) | 682.6 (277.5)
Hoehn & Yahr Stage [Median (Inter-Quartile Range); unit: Stage] — The Modified Hoehn & Yahr Scale is a standard staging system for Parkinson disease, defined by motor function. Stages are as follows:
  1. Unilateral involvement only 1.5: Unilateral and axial involvement
  2. Bilateral involvement without impairment of balance 2.5: Mild bilateral disease with recovery on pull test
  3. Mild to moderate bilateral disease with some postural instability but physically independent
  4. Severe disability; still able to walk or stand unassisted
  5. Wheelchair-bound or bedridden unless aided. Only subjects in stages 1-3 were included in the study.
  Stage | 2 [2 to 2] | 2 [2 to 2] | 2 [2 to 2]
MDS-UPDRS Part 3 Score [Median (Inter-Quartile Range); unit: units on a scale] — The Movement Disorder Society's Unified Parkinson's Disease Rating Scale (MDS-UPDRS) is a validated, comprehensive scale commonly used to rate the severity of signs (Part 3) and symptoms (Parts 1, 2, and 4) in Parkinson's Disease. In all parts, higher scores indicate more severe symptoms/signs and greater disability. Part 1 rates non-motor symptoms with scores ranging 0-52. Part 2 rates motor symptoms again 0-52. Part 3 rates motor signs, as evaluated by a trained clinician, with scores 0-132. Part 4 rates motor complications 0-24. Here, only Part 3 is used as a measure of PD motor severity.
  units on a scale | 24 [20 to 28] | 24.5 [21 to 34] | 24 [20 to 30]

OUTCOME MEASURES:

1. Primary Outcome: Change in Sleep Efficiency as Measured by Polysomnogram
Description: Sleep efficiency is defined as total sleep time divided by total time in bed, expressed as a percent. Polysomnograms were performed at baseline, end of treatment period 1, and end of treatment period 2. A positive change indicates improvement in sleep efficiency. Assessing difference between change in sleep efficiency during suvorexant period and change in sleep efficiency during placebo period.
Time Frame: 4 weeks
Measure: Median (Inter-Quartile Range); unit: Percentage (see sleep efficiency def)
Groups:
- Suvorexant Period: All subjects assessed during suvorexant period, regardless of whether they received suvorexant in treatment period 1 or treatment period 2.
- Placebo: All Subjects assessed during placebo treatment, regardless of whether this was treatment period 1 or treatment period 2
Arm/Group | Suvorexant Period | Placebo
Number analyzed (Participants) | 19 | 19
Percentage (see sleep efficiency def) | 8.9 [-3.1 to 14.5] | 9.4 [3.2 to 13.6]
Statistical Analysis 1: Comparison: Suvorexant Period vs Placebo; Test type: Superiority; p = 0.72, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Wakefulness After Sleep Onset (WASO)
Description: Wakefulness after sleep onset (WASO) is defined as total time spent awake after first epoch of sleep and before final awakening. Captured during polysomnograms performed at baseline, end of treatment period 1, and end of treatment period 2. Measured in minutes. A negative change indicates improvement in WASO.
Time Frame: 4 weeks
Measure: Median (Inter-Quartile Range); unit: Minutes
Groups:
- Suvorexant: All subjects assessed during suvorexant period, regardless of whether they received suvorexant in treatment period 1 or treatment period 2.
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 19 | 19
Minutes | -54.1 [-61.0 to 22.5] | -36.5 [-54.0 to 0.0]
Statistical Analysis 1: Comparison: Suvorexant vs Placebo; Test type: Superiority; p = 0.51, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Latency to Persistent Sleep (LPS)
Description: Latency to Persistent Sleep (LPS) is defined as total time between lights out and first epoch of sleep. Measured on polysomnogram performed at baseline, end of treatment period 1, and end of treatment period 2. A negative change indicates improvement in LPS.
Time Frame: 4 weeks
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 19 | 19
Minutes | -9.4 [-26.1 to 1.3] | -4.2 [-11.2 to 0.0]
Statistical Analysis 1: Comparison: Suvorexant vs Placebo; Test type: Superiority; p = 0.81, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Insomnia Severity Index (ISI)
Description: The Insomnia Severity Index (ISI) is a 7-question survey assessing symptoms of insomnia. Scores range from 0 to 28, with higher scores indicating greater severity. Thus, a negative change in the ISI score indicates improvement in sleep. Performed at baseline, end of treatment period 1, start of treatment period 2, and end of treatment period 2.
Time Frame: 4 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 19 | 19
units on a scale | -1 [-4 to 0] | 1 [-0.5 to 3.5]
Statistical Analysis 1: Comparison: Suvorexant vs Placebo; Test type: Superiority; p = 0.004, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Epworth Sleepiness Scale (ESS)
Description: The Epworth Sleepiness Scale (ESS) is an 8-question survey assessing symptoms of daytime sleepiness. Scores range from 0 to 24, with higher scores indicating greater severity of daytime sleepiness. Thus, a negative change indicates improvement in daytime sleepiness. The ESS has been validated for use in the general population and in PD. Administered at start of treatment period 1, end of treatment period 1, start of treatment period 2, and end of treatment period 2.
Time Frame: 4 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 19 | 19
units on a scale | -0.5 [-3.0 to 1.0] | 0.0 [-1.0 to 2.0]
Statistical Analysis 1: Comparison: Suvorexant vs Placebo; Test type: Superiority; p = 0.32, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Subject's Global Impression of Change (SGI-C)
Description: The Subject's Global Impression of Change (SGI-C) is a rating scale that asks a single question: "Since baseline (when first starting this study), how have your sleep symptoms changed?" Answers will be on a 7-point scale: 1 = much improved; 2 = somewhat improved; 3 = minimally improved; 4 = no change; 5 = minimally worse; 6 = somewhat worse; and 7 = much worse. Evaluated at end of treatment period 1 and end of treatment period 2.
Time Frame: 4 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 19 | 19
score on a scale | 3 [2 to 4] | 4 [3 to 4]
Statistical Analysis 1: Comparison: Suvorexant vs Placebo; Test type: Superiority; p = 0.098, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Clinician's Global Impression of Change (CGI-C)
Description: The Clinician's Global Impression of Change (CGI-C) is a rating scale that asks the single question: "Since baseline (when first starting this study), how have the subject's sleep symptoms changed?" Answers will be on a 7-point scale: 1 = much improved; 2 = somewhat improved; 3 = minimally improved; 4 = no change; 5 = minimally worse; 6 = somewhat worse; and 7 = much worse.
Time Frame: 4 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 19 | 19
score on a scale | 3 [2 to 4] | 4 [3 to 4]
Statistical Analysis 1: Comparison: Suvorexant vs Placebo; Test type: Superiority; p = 0.2, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse event data for each subject was recorded over the duration of their participation in the study, which was 11-15 weeks.
Arm/Group | Suvorexant | Placebo
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 2/21 | 3/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Suvorexant (N=21) | Placebo (N=21)
Excessive Drowsiness (Nervous system disorders) | 2 | 2
Nausea (Gastrointestinal disorders) | 0 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 0
Compulsive behavior (Nervous system disorders) | 0 | 1 (2)

LIMITATIONS AND CAVEATS:
Designed as a pilot study, so recruitment goal was low and consequently the sample size is small, limiting interpretation of the significance of the differences between suvorexant and placebo.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-08): https://cdn.clinicaltrials.gov/large-docs/14/NCT02729714/Prot_SAP_000.pdf